CLINICAL TRIAL: NCT03426163
Title: Effect of Preoperative MRI Virtual Reality in Patients Undergoing Knee: a Randomized Controlled Trial
Brief Title: Effect of Preoperative MRI Virtual Reality in Patients Undergoing Knee Arthroscope Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanyang University Seoul Hospital (Other)
Responsible Party: Principal Investigator, JIN KYU LEE, Assistant Professor, Hanyang University Seoul Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Hanyang University
Record Dates: First submitted 2018-01-29; First posted 2018-02-08 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Knee Injuries
Keywords: virtual reality; knee
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR group (Experimental): Application of virtual reality 12 hours before arthroscopic surgery
  Interventions: Device: Virtual reality
- Non-VR group (No Intervention): Application of knee MRI 12 hours before arthroscopic surgery

INTERVENTIONS:
Device: Virtual reality — Application of knee MRI transformed virtual reality system
  Arms: VR group

SUMMARY:
Knee MRI is difficult for patients to understand as the image offers a single plane image. Accordingly,investigators sought to transfer the MRI image to 3-dimensional virtual reality system by Mesh rendering technique.

DETAILED DESCRIPTION:
The primary outcome of the study is APAIS score assessed at 24 hours postoperation. Experimental VR group will be applied with virtual reality transformed knee MRI whereas no interverntion group will be applied with traditional knee MRI. MRI will be transformed to virtual reality images by Mesh rendering technique.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective knee arthroscopy surgery

Exclusion Criteria:

* Infection, not willing to undergo study, mentally ill, severe osteoarthritis (KL grade III or more)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-06-15 (Estimated); Study Completion 2018-08-15 (Estimated)

PRIMARY OUTCOMES:
The Amsterdam perioperative anxiety and information scale (APAIS) score | postoperatively at 24 hours
  surgery related anxiety and information score
  Interpretation:
  * minimum subscale scores: 2
  * minimum combined anxiety component: 4
  * maximum subscale scores: 10
  * maximum combined anxiety component: 20
  * The higher the scores the greater the degree of anxiety or need for additional information.

SECONDARY OUTCOMES:
Visual analogue scale (VAS) for satisfaction | postoperatively at 24 hours
  Satisfaction scale with a range of scores from 0-100. A higher score indicates greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: JIN KYU M LEE, Study Chair — Hanyang University Seoul Hospital
Locations (1):
- Hanyang University Seoul Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang JH, Ryu JJ, Nam E, Lee HS, Lee JK. Effects of Preoperative Virtual Reality Magnetic Resonance Imaging on Preoperative Anxiety in Patients Undergoing Arthroscopic Knee Surgery: A Randomized Controlled Study. Arthroscopy. 2019 Aug;35(8):2394-2399. doi: 10.1016/j.arthro.2019.02.037. PMID 31395176